CLINICAL TRIAL: NCT02866682
Title: Prospective Study Comparing Brand and Generic Immunosuppression on Transplant Outcomes, Adherence, & Immune Response
Brief Title: Prospective Study Comparing Brand and Generic Immunosuppression on Transplant Outcomes, Adherence, & Immune Response in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Suphamai Bunnapradist, Professor of Medicine, Director of Research, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-001423
Record Dates: First submitted 2016-07-26; First posted 2016-08-15 (Estimated); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Renal Transplant Rejection
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brand Tacrolimus Only : Prograf (Other): Arm 1 will receive brand tacrolimus for the entire study
  Interventions: Drug: Prograf
- Generic A Only (Other): Arm 2 will receive specific generic tacrolimus for the entire study
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Prograf — Brand Drug for the duration of the study.
  Arms: Brand Tacrolimus Only : Prograf
Drug: Tacrolimus — Generic
  Arms: Generic A Only

SUMMARY:
As the patents for brand-name immunosuppressive medications expire, there is increasing interest in using generic immunosuppressive drugs. However, despite pharmacokinetic studies showing bioequivalence, questions remain regarding the clinical impact of use of generic immunosuppression.

The most important immunosuppressive agent in the modern transplant era is arguably tacrolimus, a calcineurin-inhibitor with a narrow therapeutic index. This study seeks to answer the question regarding the clinical impact of generic tacrolimus use as measured primarily by acute rejection, loss of graft function, and patient death through a randomized trial of 2 phases: Brand tacrolimus only, and Generic A tacrolimus only. Given that kidney transplantations are the most commonly performed transplants with well-defined measures of rejection and graft failure, this organs will be studied in a six-center study designed to accrue the target number of transplant recipients within the one-year study period.

The study has now been branched off into 2 phases. Phase 1: consists of randomization of patients onto brand and generic tacrolimus. This was completed once 40 brand patients were enrolled. Phase 2: consists of patients being enrolled only on generic tacrolimus (standard of care from subject's insurance). This will be completed once there is a total of 160 generic participants. 200 participants total in the study.

DETAILED DESCRIPTION:
A prospective, randomized, open-label, multicenter, parallel, observational study to assess safety and efficacy of 200 kidney transplant recipients comparing brand tacrolimus to generic tacrolimus over a one year follow up period. All subjects will receive other immunosuppressive medications including induction therapy (thymoglobulin, basiliximab, or no induction) and maintenance including mycophenolate mofetil and corticosteroid therapy as directed by standard-of-care at each center. Their medication information will be recorded in their study files.

The study population includes recipients of kidney allografts in the first 14 days after transplantation.

The totals of 7 visits over 12 months period are planned as follows. The blood samples specified below are for the translational research study labs. Subjects will continue to receive routine labs as part of their standard of care from their treating physician. These safety labs are done as part of their stand of care from their treating physician.

If the subject needs more study drug medication before his or her next study visit the subject will come in to the clinic to get a new supply.

First (Baseline) Visit (up to 14 days after transplant but before you are discharged from the hospital):

* Review and sign this consent form
* Review of your medical history
* Review of your current medications
* Review of your physical exam including vital signs (blood pressure, temperature, pulse and respiration rate), height and weight
* Review of clinical labs
* You will receive your study drug if you are in Part 1 of the study.

If you are a woman of child bearing potential, a pregnancy test will be completed prior to the start of the study. If you are pregnant, you cannot participate in this research study. You also cannot participate in this study if you are currently breastfeeding. You must use a medically acceptable method of birth control during the 1-year study period and for 6 weeks after the last dose of study medication.

It is possible that after the study doctor reviews your medical history and test results, he or she may tell you that you do not qualify to be in the study. If you do not qualify for the study, the doctor will tell you the reason(s) why. If you cannot be in this research study, you will not lose any medical benefits, you can still participate in other studies, and you can still receive the standard treatment prescribed by your physician.

After the Baseline Visit, you will have 6 additional study visits. These will be scheduled for 1, 2, 3, 6, 9, and 12 months after your transplant surgery. The following will occur at each visit:

Month 1, 2, 3, 6, and 9 Visits:

* Review of your current medications
* Review of your physical exam including vital signs (blood pressure, temperature, pulse and respiration rate), height and weight
* Review of any changes in your health and any reactions to the study medication will be recorded
* Review of your routine standard of care lab results
* Return completed dosing diary and receive new dosing diary
* You will receive your study drug if you are in Part 1 of the study

Month 12 Visit (End of Study Visit):

* Review of your current medications
* Review of any changes in your health and any reactions to the study medication will be recorded
* Review of your routine standard of care lab result
* Return your final completed dosing diary
* Return any study drug remaining in your possession to the study team if you are in Part 1 of the study

If you are Part 1 and require more study medication before your next study visit, you will come in to the clinic to get a new supply. If you are participating in Part 2, you will obtain more study drug from your local pharmacy.

You will continue having your routine blood and urine collections to monitor your kidney function as part of your standard of care treatment at UCLA, UCSD, UCI, and UCD. The schedule for these routine blood and urine collections will depend on your condition and will be at your treating physician's discretion.

Adherence will be measured with daily medication diaries and with the coefficient of variation of tacrolimus in subjects' blood.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent and or/assent
2. Between the ages of 18 and 70 years, inclusive
3. Current or future kidney transplant recipients, no more than 14 days after transplant and prior to hospital discharge. Inclusion of future kidney transplant recipients cannot exceed 30-days pre-transplant.
4. Able to swallow tablets and capsules at the time of randomization
5. Subjects must be receiving a primary or secondary kidney allograft from a deceased donor or from a non- HLA identical living donor
6. Negative cross match test, and compatible (A, B, AB or O) blood type
7. Subjects must have no known contraindications to tacrolimus
8. Women of childbearing potential (WOCBP) must have a negative pregnancy test and be willing to use 2 methods of contraception during the study and for 6 weeks after stopping the study drug.

WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone level > 35 mIU/cc). Women who are using oral, implanted, or injectable contraceptive hormones (intrauterine device), mechanical products or barrier methods (diaphragm, condoms, spermicides), are practicing abstinence, or have a sterile partner (e.g., vasectomy), will be considered of child bearing potential.

In addition, WOCBP who are taking MMF must use methods of birth control as stipulated in the package insert, namely:

Either intrauterine device, or partner with vasectomy, or one hormone (oral contraceptive pill, transdermal patch, vaginal ring, or progesterone injection or implant) and one barrier method (diaphragm or cervical cap with spermicide, contraceptive sponge, or male or female condom), or two barrier methods as described above.

WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at the time of transplant.

Exclusion Criteria

1. Those who receive simultaneous combined organ transplants
2. Subjects with clinically significant active infections (for example, those requiring hospitalization, or as judged by the Investigator) or malignancies
3. Recipients who are concurrently receiving belatacept or anticipate to receive belatacept as part of their immunosuppressive regimen
4. Subjects currently enrolled in another investigational device or drug study
5. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for 6 weeks after stopping the study drug
6. Women who are breast-feeding or pregnant with a positive pregnancy test on enrollment or prior to study drug administration
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
8. Any psychiatric or medical condition that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suphamai Bunnapradist, M.D.,M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Kidney Transplant Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants withdrew prior to randomization.
Period: Overall Study
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Started | 39 | 132
Completed | 39 | 120
Not Completed | 0 | 12
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 4
Not completed — Tacrolimus Discontinued During Study | 0 | 6
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only | Total
Number analyzed (Participants) | 39 | 132 | 171
Age, Continuous [Median (Standard Deviation); unit: years] | 53.0 (12.7) | 52.2 (13.1) | 52.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 58 | 73
  Male | 24 | 74 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 9 | 33 | 42
  Black | 5 | 12 | 17
  Asian | 3 | 12 | 15
  Hispanic or Latino | 12 | 50 | 62
  Multiracial | 6 | 25 | 31
  American Indian or Alaska Native | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 132 | 171

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Acute Rejection, Failure, Death
Description: The definition of graft failure includes re-transplant and/or death and, in case of kidney transplant, also includes return to dialysis. Acute rejection was defined as biopsy-proven rejection according to Banff 2007 criteria. Please see the following article for details of the Banff '07 classification: https://www.sciencedirect.com/science/article/pii/S1600613522056428?via%3Dihub.
Time Frame: 1 year post-transplant
Population: No participants experienced graft rejection or death in the Brand Tacrolimus group. Only 1 participant on the Brand group experienced graft failure. On the other hand, the generic group had 9 participants that experienced rejection, 1 that experienced graft failure, and 1 that experienced death.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 1 | 11
days
  Time to first of rejection: number analyzed (Participants) | 0 | 9
  Time to first of rejection |  | 57.1 (66.5)
  Time to first graft failure: number analyzed (Participants) | 1 | 1
  Time to first graft failure | 86 | 200
  Time to first death: number analyzed (Participants) | 0 | 1
  Time to first death |  | 200

2. Secondary Outcome: Number of Participants With Graft Rejection at 1 Year
Description: Rejection was defined as biopsy-proven rejection according to Banff 2007 criteria. Please see the following article for details of the Banff '07 classification: https://www.sciencedirect.com/science/article/pii/S1600613522056428?via%3Dihub.
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 39 | 120
Participants | 0 | 9

3. Secondary Outcome: Number of Participants With Graft Failure at 1 Year
Description: Graft failure as determined by return to dialysis, death, or re-transplant
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 39 | 120
Participants | 1 | 1

4. Secondary Outcome: Number of Participants With Infectious Episodes at 1 Year
Description: Infectious episodes are defined as a positive test result for an infection.
Time Frame: 1 year post-transplant
Measure: Number; unit: participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 39 | 120
participants
  Cytomegalovirus infection | 10 | 22
  BK virus infection | 3 | 16
  Other infection | 15 | 34

5. Secondary Outcome: Number of Participants With Malignancy at 1 Year
Description: Malignancy is defined as physician reported malignancy according to review of participants' medical history.
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 39 | 132
Participants | 0 | 1

6. Secondary Outcome: Death or Loss-to-follow-up at 1 Year
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 39 | 132
Participants | 0 | 5

7. Secondary Outcome: Changes in Lymphocyte Subpopulations and Production of Donor Specific HLA Antibodies
Time Frame: post-transplant
Population: Outcome was not collected or measured due to approved changes in protocol amendment
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Adhered to Medication Regimen
Description: Patient adherence was assessed by their physician with participants marked as "adherent," "non-adherent," or "unknown."
Time Frame: post-transplant
Population: Remaining participants did not have adherence data collected due to appointment cancellations during Covid-19 pandemic
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 37 | 106
Participants | 37 | 105

9. Secondary Outcome: Quality of Life With Medication Regimen
Time Frame: post-transplant
Population: This was not collected due to protocol amendment changes which no longer required this outcome data.
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Satisfaction With Medication Regimen
Time Frame: post-transplant
Population: Outcome not measured or collected due to approved changes in protocol amendment
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year Post-Transplant
Arm/Group | Brand Tacrolimus Only : Prograf | Generic A Only
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/132
Serious Adverse Events (participants affected / at risk) | 19/39 | 43/132
Other Adverse Events (participants affected / at risk) | 32/39 | 105/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brand Tacrolimus Only : Prograf (N=39) | Generic A Only (N=132)
Life threatening event associated with an immediate risk of death (General disorders) | 0 (0) | 1 (1)
Re-hospitalization (General disorders) | 13 (30) | 41 (98)
Prolonged hospitalization (General disorders) | 10 (15) | 6 (6)
Important medical event requiring medical intervention (General disorders) | 1 (1) | 1 (1) — The patient had an important medical event that, based upon the investigator's medical judgment, may significantly jeopardize the patient's health and require medical or surgical intervention to prevent negative outcomes
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brand Tacrolimus Only : Prograf (N=39) | Generic A Only (N=132)
Abdominal Pain (Gastrointestinal disorders) | 6 | 14
Acute Kidney Injury (Renal and urinary disorders) | 9 | 30
Anemia (Blood and lymphatic system disorders) | 6 | 33
Constipation (Gastrointestinal disorders) | 5 | 17
Diarrhea (Gastrointestinal disorders) | 11 | 27
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 9
Hematuria (Renal and urinary disorders) | 5 | 10
Hypercalcemia (Metabolism and nutrition disorders) | 13 | 20
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 21
Hyperkalemia (Metabolism and nutrition disorders) | 14 | 41
Hyperphosphatemia (Metabolism and nutrition disorders) | 7 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 14
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hypomagnesimia (Metabolism and nutrition disorders) | 14 | 59
Hypophosphatemia (Metabolism and nutrition disorders) | 12 | 51
Hypotension (Cardiac disorders) | 4 | 10
Impaired Fasting Blood Glucose (Metabolism and nutrition disorders) | 8 | 6
Incisional Pain (Injury, poisoning and procedural complications) | 5 | 7
Infection (Infections and infestations) | 20 | 55
Leukocytosis (Immune system disorders) | 7 | 15
Leukopenia (Immune system disorders) | 12 | 41
Lower extremity edema (Renal and urinary disorders) | 6 | 6
Metabolic Acidosis (Metabolism and nutrition disorders) | 12 | 29
Nausea (Gastrointestinal disorders) | 4 | 16
Neutropenia (Immune system disorders) | 5 | 6
Post Operative Pain (Injury, poisoning and procedural complications) | 0 | 19
Pyuria (Renal and urinary disorders) | 9 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 8
Transaminitis (Hepatobiliary disorders) | 9 | 27
Tremor (Musculoskeletal and connective tissue disorders) | 5 | 24
Abnormal Urinalysis (Renal and urinary disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Deep Vein Thrombosis (Vascular disorders) | 2 | 4
de novo DSA (Immune system disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Edema (General disorders) | 1 | 7
Fatigue (General disorders) | 2 | 3
Headache (General disorders) | 3 | 5
Hypertension (Cardiac disorders) | 1 | 11
Elevated BUN (Renal and urinary disorders) | 2 | 0
Kidney Transplant Rejection (Renal and urinary disorders) | 0 | 9
Orthostatic Hypotension (Cardiac disorders) | 0 | 8
Proteinuria (Renal and urinary disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 9
Secondary Hyperparathyroidism (Endocrine disorders) | 2 | 0
Uncontrolled Diabetes (Endocrine disorders) | 2 | 1
Vomiting (General disorders) | 3 | 5
Weight Gain (General disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02866682/Prot_SAP_000.pdf